CLINICAL TRIAL: NCT03684421
Title: Clinical and Live Birth Rates After Controlled Ovarian Stimulation With the Long Antagonist Protocol Versus Classical Antagonist Protocol
Brief Title: Clinical and Live Birth Rates After Following Long Antagonist Protocol Versus Classical Antagonist Protocol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assisting Nature (Other)
Responsible Party: Principal Investigator, Papanikolaou Evaggelos, Papanikolaou Evaggelos, MD, PhD, Assisting Nature
Other Study IDs: Long-Ant-vs-Ant-AN006
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pregnancy, Ovarian
Keywords: Long Antagonist; Classical Antagonist; live birth rate; clinical pregnancy rate; ovarian stimulation; IVF
MeSH Terms: conditions — Pregnancy, Ovarian | interventions — Pregnancy Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long Antagonist Protocol: Clinical pregnancy rate and live birth rates of patients who followed Long Antagonist Protocol for COS
  Interventions: Diagnostic Test: Pregnancy Rate
- Classical Antagonist Protocol: Clinical pregnancy rate and live birth rates of patients who followed Classical Antagonist Protocol for COS
  Interventions: Diagnostic Test: Pregnancy Rate

INTERVENTIONS:
Diagnostic Test: Pregnancy Rate — The clinical pregnancy and live birth rate according to the protocol of COS

SUMMARY:
A randomized prospective study of the evaluation of the clinical IVF results after following Long Antagonist protocol for controlled ovarian stimulation versus following classical antagonist protocol

DETAILED DESCRIPTION:
A randomized prospective study of administration of Degarelix in late luteal phase of women undergoing ovarian stimulation for IVF: Single dose of Degarelix (24mg, 16mg or 12 mg), on day 24th of previous luteal face cycle, was administered. The Clinical Pregnancy and Live Birth Rates were estimated for this group of patients, comparing to the rates of the group which followed classical antagonist protocol. The number of the formed blastocysts in each group is measured, as well.

ELIGIBILITY:
Inclusion Criteria:

* primary infertility
* age 18-39 years; body mass index (BMI) 18-29kg/m2;
* regular menstrual cycle of 26-35days,
* presumed to be ovulatory;
* early follicular- phase serum concentration of FSH within normal limits (1-12 IU/l).

Exclusion Criteria:

* women with diabetes and other metabolic disease
* women with heart disease, QT prolongation,heart failure
* elevated liver enzymes, liver failure, hepatitis
* women with inflammatory or autoimmune disease
* abnormal karyotype;
* polycystic ovarian syndrome,
* endometriosis stage III/IV;
* history of being a 'poor responder',
* defined as >20 days of gonadotrophin in a previous stimulation cycle, or any previous cancellation of a stimulation cycle due to limited follicular response, or development of less than 4 follicles 15 mm in a previous stimulation cycle; history of recurrent miscarriage; severe OHSS in a previous stimula- tion cycle or any contraindication for the use of gonadotrophins.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women 18- 39 years old who follow COS with the Long Antagonist Protocol or with Long Agonist Protocol
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate according to stimulation protocol | 6 weeks to 42 weeks after embryo transfer
  Clinical Pregnancy Rate according to stimulation protocol
Number of formed blastocysts | 5 days after the OPU day
  The number of the formed blastocysts in each group

SECONDARY OUTCOMES:
Live Birth Rate according to stimulation protocol | 6 weeks to 42 weeks after embryo transfer
  Live Birth Rate according to stimulation protocol

CONTACTS AND LOCATIONS:
Overall Officials: Evaggelos Papanikolaou, MD, PhD, Principal Investigator — Assisting Nature; Robert Najdecki, MD, PhD, Principal Investigator — Assisting Nature
Locations (1):
- Assisting Nature, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided